CLINICAL TRIAL: NCT02406443
Title: Effects of DPP-4 Inhibitor Therapy on Renal Sodium Handling and Renal Hemodynamics in Type 2 Diabetes Patients. The INDORSE Study: Inhibition of Dipeptidyl Peptidase IV: Outcomes on Renal Sodium Excretion
Brief Title: The INDORSE Study: Inhibition of Dipeptidyl Peptidase IV: Outcomes on Renal Sodium Excretion
Acronym: INDORSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14-8616
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes, DPP-4 inhibitors, renal sodium excretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): sitagliptin (DPP-4 inhibitor) oral tablet (100 mg); Januvia; administered once daily for 28 days
  Interventions: Drug: Sitaglitpin
- Placebo arm (Placebo Comparator): placebo (no medicinal ingredients) oral tablet (100 mg); administered once daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sitaglitpin — Oral DPP-4 inhibitor, 100 mg tablet administered once daily for 28 days
  Other Names: Januvia
  Arms: Experimental arm
Other: Placebo — Oral tablet (no medicinal ingredients) administered once daily for 28 days
  Arms: Placebo arm

SUMMARY:
Background: Dedicated renal hemodynamic and renal function studies are lacking for DPP-4 inhibitors in patients with Type 2 diabetes; accordingly little is known regarding the mechanisms mediating the renal effects of DPP-4 inhibitors in humans.

Objectives: To evaluate the effect of DPP-4 inhibition acutely (single dose) and following short-term therapy (28 days) on renal sodium handling and renal hemodynamics and function in patients with type 2 diabetes and systolic hypertension.

Design: double-blind, randomized, placebo-controlled trial, Phase IV.

Patient population: 32 patients with Type 2 diabetes, HbA1c (6.5%-9%), with systolic blood pressure ranging from 120-160 mmHg.

Intervention: subjects will be randomized (1:1) to either sitagliptin (100 mg daily) or to placebo (1 tablet daily) for 28 days.

Endpoints: Fractional excretion of sodium, renal function, and renal hemodynamics.

DETAILED DESCRIPTION:
Background: DPP-4 inhibition improves glycemic control, modestly reduces blood pressure and may also reduce albuminuria in patients with Type 2 diabetes; effects which occur without significantly modifying heart rate or body weight. While preclinical studies have demonstrated that DPP-4 inhibition acutely increases urinary sodium excretion in addition to other favorable renal effects (anti-inflammatory, anti-proteinuric), few studies have examined the renal effects of DPP-4 inhibition either acutely or following short-term therapy in humans with type 2 diabetes. Considering the world-wide prevalence of Type 2 diabetes and the increasing use of DPP-4 inhibitors amongst patients, it is important to ascertain potential non-glycemic effects of DPP-4 inhibitors including those within the kidney.

Study Objectives: To determine effect(s) of DPP-4 inhibition on tubular sodium handling, renal hemodynamics, and renal function.

Study Design: double-blind, randomized, placebo-controlled trial, Phase IV.

Study Patients: 32 patients with Type 2 Diabetes and Systolic Hypertension (SBP 120-160 mmHg).

Endpoints: Fractional excretion of sodium, renal function (measured GFR), renal hemodynamics (effective renal plasma flow, filtration fraction, renal blood flow, renal vascular resistance), systemic hemodynamics (non-invasive cardiac monitoring), plasma neurohormones, urinary vasoactive mediators, markers of free radical stress.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18-70 years of age,
* with Type 2 Diabetes,
* with an HbA1c (6.5%-9%),
* and with a systolic blood pressure (120-160 mmHg).

Exclusion Criteria:

* Individuals with:

  1. Type 1 Diabetes,
  2. eGFR <50mL/min/1.73m,
  3. pregnancy or breast feeding,
  4. significant cardiac, pulmonary or liver disease,
  5. prior history of pancreatitis, medullary thyroid cancer, multiple endocrine neoplasia syndromes,
  6. SBP >161 mmHg, 7) DBP >100 mmHg,
  7. alcohol or substance abuse,
  8. states of secondary hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovshin, MD,PhD, Study Director — Lunenfeld Tanenbaum Reserach Institute, Divsion of Endocrinology and Metabolism, University of Toronto; David I Cherney, MD,PhD, Principal Investigator — Division of Nephrology, University Health Network, University of Toronto
Locations (1):
- University Health Network - Division of Nephrology, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lovshin JA, Rajasekeran H, Lytvyn Y, Lovblom LE, Khan S, Alemu R, Locke A, Lai V, He H, Hittle L, Wang W, Drucker DJ, Cherney DZI. Dipeptidyl Peptidase 4 Inhibition Stimulates Distal Tubular Natriuresis and Increases in Circulating SDF-1alpha1-67 in Patients With Type 2 Diabetes. Diabetes Care. 2017 Aug;40(8):1073-1081. doi: 10.2337/dc17-0061. Epub 2017 May 26. PMID 28550195

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm | Placebo Arm
Started | 18 | 18
Completed | 16 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Placebo Arm | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (7.6) | 59.3 (8.8) | 59.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 11 | 9 | 20
Diabetes Duration [Median (Inter-Quartile Range); unit: years] | 6.0 [3.0 to 10.0] | 8.5 [5.5 to 14.0] | 8.0 [4.0 to 10.0]
HbA1c (%) [Mean (Standard Deviation); unit: Percentage] | 7.18 (0.97) | 7.31 (0.84) | 7.2 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fractional Excretion of Sodium (FENA)
Description: FENA at 3Hrs post-study drug administration after 1 month compared to FENA at 3Hrs post-study drug administration after 1 dose expressed as percent change, sitagliptin vs. placebo
Time Frame: 3 Hrs post-administration after 1 month and after 1 dose
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
percentage of change | 41 (43) | -5.0 (31)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p = 0.012, Regression, Linear; Mean Difference (Final Values) = 46

2. Secondary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: Measured GFR (Inulin Clearance) at 3Hrs post study-drug after 1 month compared to Measured GFR at 3Hrs post-study drug after 1 dose, sitagliptin vs. placebo
Time Frame: 3 Hrs post-administration after 1 month and after 1 dose
Measure: Mean (Standard Deviation); unit: ml per min per 1.73 m2
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
ml per min per 1.73 m2 | 3.9 (20.4) | -1.8 (17.8)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p = 0.40, Regression, Linear; Median Difference (Final Values) = 5.7

3. Secondary Outcome: Change in Fractional Excretion of Lithium (FELi)
Description: FELi at 3 Hr post-study drug administration after 1 month compared to FELI at 3hrs post-study drug administration after 1 dose, sitagliptin vs. placebo
Time Frame: 3 Hrs post-administration after 1 month and after 1 dose
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
percentage of change | 29 (55) | 7 (44)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Final Values) = 22

4. Secondary Outcome: Change From Baseline in SDF-1alpha^1-67 (Intact) Measured by Immunoaffinity and Tandem Mass Spectrometry
Description: Plasma concentration of SDF-1alpha^1-67 (intact) measured by quantitative mass spectrometry methods after antibody-based affinity enrichment, sitagliptin vs. placebo
Time Frame: 3 Hr vs. baseline after 1 dose
Measure: Mean (Standard Deviation); unit: ng per mL
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
ng per mL | 0.5 (0.2) | 0 (0)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 0.5

5. Secondary Outcome: Change From Baseline in SDF-1alpha^3-67 (Truncated) Measured by Tandem Mass Spectrometry With Antibody-based Affinity Enrichment
Description: Plasma concentration of SDF-1alpha^3-67 (intact) measured by quantitative mass spectrometry methods after antibody-based affinity enrichment, sitagliptin vs. placebo
Time Frame: 3Hrs vs baseline after 1 dose
Measure: Mean (Standard Deviation); unit: ng per mL
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
ng per mL | -2.0 (0.4) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 2.4

6. Secondary Outcome: Change in Systolic Blood Pressure (SBP), Non-invasive Cardiac Output Monitoring
Description: SBP by Non-Invasive cardiac output monitoring at 3Hrs post- study drug administration after 1 month compared to SBP by Non-invasive cardiac output monitoring at 3Hrs after 1 dose, sitagliptin vs placebo
Time Frame: 3 Hrs post-administration after 1 month and after 1 dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
mmHg | 5.7 (9.9) | 0.0 (14.0)
Statistical Analysis 1: Comparison: Experimental Arm vs Placebo Arm; Test type: Superiority; p = 0.42, Regression, Linear; Mean Difference (Final Values) = 5.7

7. Secondary Outcome: Change in Effective Renal Plasma Flow (ERPF)
Description: ERPF (para-aminohippurate clearance) 3Hrs post-study drug administration after 1 month compared to ERPF at 3Hhrs post-study drug administration after 1 dose, sitagliptin vs placebo
Time Frame: 3 Hrs post-administration after 1 month and after 1 dose
Measure: Mean (Standard Deviation); unit: ml per min per 1.73 m2
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 16 | 16
ml per min per 1.73 m2 | 31.1 (152.1) | -24.7 (142.8)

ADVERSE EVENTS:
Description: The intention to treat population at risk was 17 for the experimental arm and 18 for the placebo arm, and the final per-protocol population was 16 per arm. 1 participant in the experimental arm was withdrawn due to lower GI bleeding after randomization, and 2 participants in the placebo arm were withdrawn, 1 due to dyspnea and 1 due to presyncope after randomization.
Arm/Group | Experimental Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=17) | Placebo Arm (N=18)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1)
Lower GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No